CLINICAL TRIAL: NCT00947505
Title: A Randomized, Double-Blind, Control Device Clinical Trial to Evaluate the Safety and Efficacy of the HairMax LaserComb 2009, 7 Beam Model: For the Treatment of Androgenetic Alopecia in Males
Brief Title: Treatment of Androgenetic Alopecia in Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lexington International, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7 2009-M-01
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Androgenetic Alopecia; Hair Loss; Male Pattern Baldness
Keywords: Androgenetic alopecia; Hair loss; Male Pattern baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HairMax LaserComb 2009, 7 Beam (Active Comparator): Lower level laser phototherapy medical device with 7 laser beams
  Interventions: Device: HairMax LaserComb 2009, 7 Beam
- Control Device (Active Comparator): Identical to the Active device, but with 7 LED's instead of lasers
  Interventions: Device: HairMax LaserComb

INTERVENTIONS:
Device: HairMax LaserComb 2009, 7 Beam — Device application 3 times week (non-consecutive days), for 26 weeks
  Other Names: HairMax LaserComb
  Arms: HairMax LaserComb 2009, 7 Beam
Device: HairMax LaserComb — Device application 3 times week (non-consecutive days), for 26 weeks
  Other Names: Control device
  Arms: Control Device

SUMMARY:
The purpose of this study is to evaluate the efficacy of the HairMax LaserComb 2009 7 Beam model in promoting hair growth in males diagnosed with androgenetic alopecia when treatment is applied as directed.

DETAILED DESCRIPTION:
This is randomized, double-blind, control device clinical study across 2 sites, evaluating changes in terminal hair-count in the evaluation zone having evidence of androgenetic alopecia (miniaturized hair).

The trial will involve 45 male subjects who have been diagnosed with androgenetic alopecia, who are between 25 and 60 years of age, have Fitzpatrick Skin Types I-IV, with classifications of Norwood-Hamilton IIa to V, have active hair loss within the last 12 months.

Subjects will use the device on three nonconcurring days a week as directed per device for 26 weeks treatment duration.

Initial efficacy endpoint for each subject will be assessed at visit 4 (week 16).

Safety analysis will be assessed based on the reports of adverse events during study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of androgenetic alopecia
* Fitzpatrick Skin Types I-IV
* Norwood-Hamilton IIa to V
* Active hair loss within last 12 months

Exclusion Criteria:

* Photosensitivity to laser light
* Malignancy in the target area

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jarratt, M.D., Principal Investigator — DermaResearch, Inc.; Abe Marcadis, M.D., Principal Investigator — Palm Beach Research Center
Locations (2):
- United States (2):
  - Abe Marcadis, M.D., Palm Beach, Florida
  - Michael Jarratt, MD, Austin, Texas

REFERENCES:
- [Background] Leavitt M, Charles G, Heyman E, Michaels D. HairMax LaserComb laser phototherapy device in the treatment of male androgenetic alopecia: A randomized, double-blind, sham device-controlled, multicentre trial. Clin Drug Investig. 2009;29(5):283-92. doi: 10.2165/00044011-200929050-00001. PMID 19366270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male subjects who have been diagnosed with androgenetic alopecia, who are between 25 and 60 years of age, have Fitzpatrick Skin Types I-Iv, with Norwood Hamilton Classifications of IIa-V, have active hair loss with the last 12 months
Pre-assignment Details: Exclusion Criteria: Individuals with photosensitivity to laser light, histor of any malignancy in target area. Also, use of phytotherapy (e.g. saw palmetto) within 8 weeks prior to baseline and use of retinoids in past year, chronic dermatological condtion (eczema , psoriasis, infection, etc.) of the scalp other than male pattern baldness
Period: Overall Study
Arm/Group | LLT Device 2009 7 Beam | Control Device
Started | 33 | 16
Completed | 24 | 14
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LLT Device 2009 7 Beam | Control Device | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 16 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 33 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Changes in Terminal Hair Count at 16 and 26 Weeks Over Baseline
Description: Results of terminal hair count will be compared to baseline for each user between active and control devicea at 26 weeks with an interim evaluation at week 16. Terminal hair count, which is non-vellus/non-miniaturized hair counts, will be assessed in the target region
Time Frame: 16 and 26 weeks
Measure: Mean (Standard Deviation); unit: change in terminal hair count
Groups:
- LLT Device 2009 7 Beam: This is the active LLLT device
- Control Device: This is the control device emitting white light
Arm/Group | LLT Device 2009 7 Beam | Control Device
Number analyzed (Participants) | 24 | 14
change in terminal hair count
  Change at 16 weeks | 17.7 (12.83) | 2.8 (6.89)
  Change at 26 weeks | 18.4 (16.6) | 1.6 (8.60)

ADVERSE EVENTS:
Arm/Group | LLT Device 2009 7 Beam | Control Device
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/14
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No